CLINICAL TRIAL: NCT02765555
Title: An Open Label, Single Center, Single Dose, Phase 1, First in Man Study of the Safety, Tolerability and Pharmacokinetic Profile of RBP-7000
Brief Title: First in Man Study of Safety, Tolerability and PK Profile of RBP-7000
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-09-0007
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RBP-7000 (Experimental): All subjects that meet initial study entry criteria will receive a test dose of 0.25mg of oral risperidone. Subjects who continue to be eligible will return to the clinical unit in one week and receive a single dose of 60mg RBP-7000 after a 2 hour fast. Subjects will remain in the clinical unit for 14 days, then return for 10 additional weeks after discharge.
  Interventions: Drug: RBP-7000

INTERVENTIONS:
Drug: RBP-7000 — Single dose

SUMMARY:
The purpose of this study is to assess the safety, tolerability and PK profile of a single dose of 60mg RBO-7000 in stable subjects with schizophrenia who are on medication other than risperidone.

DETAILED DESCRIPTION:
Twelve subjects with stable schizophrenia will be enrolled. The expected duration of participation is 88 days which includes at least a 2 days screening and an 85 day treatment period (15 -day inpatient stay in the clinical unit and an additional 70-day outpatient period, including the Day 85 end of study follow up or early termination visit. Visits will occur approximately weekly during the outpatient period.

Neurological and clinical symptom assessments (Positive and Negative Syndrome Scale [PANSS], Clinical Global Impressions-Schizophrenic Specific [CGI-SCH], Simpson-Angus Scale [SAS], Barnes Akathisia Scale [BAS], and Columbia-Suicide Severity Rating Scale [C-SSRS]) will be conducted at screening, on the day of admission to the clinical unit (Day -1), and at each post-dose visit throughout the study including the follow-up visit. Scale results will be reviewed by the Principal Investigator. The Abnormal Involuntary Movement Scale (AIMS) for Tardive Dyskinesia will be performed at screening and at each post-dose visit throughout the study including the end of study follow-up visit. CYP-2D6 genotyping will be conducted at screening. Tolerability will be measured using SAS, which will be conducted as described above.

Blood samples to assess the PK parameters will be taken from pre-dose until approximately 84 days post-dose.

End of study procedures will be conducted on follow-up Day 85 (84 days post-dose) or early termination (ET) to assess any adverse events (AEs) that were ongoing at the last visit, any new AEs that have developed, and for measurement of safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of paranoid, residual, or undifferentiated schizophrenia in a documented letter from the subject's psychiatrist or primary care provider.
* Clinically stable subjects (subjects whom the Principal Investigator (PI) established by medical record or by history from the subject and at least one reliable informant who resides with the subject, that the subject has been clinically stable for at least 60 days without hospitalization) will be eligible to participate in the study.
* Subjects with a body mass index (BMI) of 18 to 33 kg/m2 inclusive and weighing at least 49.9 kg are eligible for entry.
* Subjects who have given written informed consent.

Exclusion Criteria:

* Subjects taking any risperidone product in the last 60 days prior to study screening.
* Subjects with a history of cancer (excluding resected basal cell or squamous cell carcinoma of the skin) unless they have been disease free for ≥ 5 years.
* Subjects with another active medical condition or organ disease that may either compromise subject safety or interfere with the safety and/or outcome evaluation of the study drug. This includes, but is not limited to the following abnormalities: total bilirubin > 2.5 mg/dL (51 μmol/L), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN) or clinically significant serum creatinine > 2 x ULN, international normalized ratio (INR) ≥ 2.0. Other excluded medical conditions including, but not limited to, history of heart attack, brain injury, low blood pressure and clinically significant irregular heartbeat.
* Subjects with known diagnosis of type 1 or 2 diabetes or subjects with an abnormal Hemoglobin A1c (HbA1c) at screening.
* Subjects with clinically significant co-morbidities that could affect near-term survival.
* Subjects treated with any investigational drug within 30 days beginning study screening.
* Subjects with significant traumatic injury, major surgery or open biopsy within the past 4 weeks.
* Subjects receiving opioid or opioid-containing analgesics.
* Subjects consuming > 1 alcoholic drink per day within the last 30 days (defined as one ounce of 80 proof spirits, 12 ounces of beer, or 4 ounces of wine).
* Subjects with prior allergic reactions or sensitivities to any component of RBP-7000.
* Subjects with other concurrent uncontrolled illness that may interfere with his or her ability to participate in the trial.
* Subjects with other known contraindications or sensitivity to risperidone or other components of RBP-7000.
* Women with a positive pregnancy test at screening. Women of childbearing potential, who are pregnant or lactating, seeking pregnancy, or failing to take adequate contraceptive precautions, (e.g., an oral or injectable contraceptive, an approved hormonal implant or topical patch, an intrauterine device, abstinence. Should a female subject become sexually active, she must agree to use a double barrier method or barrier plus spermicide). A woman of childbearing potential is defined as any female who is less than 2 years post-menopausal or has not undergone a hysterectomy or surgical sterilization, e.g. bilateral tubal ligation, bilateral ovariectomy (oophorectomy).
* . Subjects with a positive urine drug screen for opiates, cocaine, amphetamines, methadone, marijuana, barbiturates, benzodiazepines, methamphetamine, phencyclidine, and tricyclic antidepressants unless the positive screen is determined to be secondary to an allowable concomitant medication.
* Subjects with epilepsy or other seizure disorders, Parkinson's disease, or dementia.
* Subjects taking buproprion, chlorpheniramine, cimetidine, clomipramine, doxepin, or quinidine.
* Subjects taking clozapine, phenothiazines, or haloperidol.
* Subjects taking serotonin reuptake inhibitors (e.g., fluoxetine, paroxetine) in the 30 days prior to beginning study screening.
* . Subjects taking medications, in addition to those listed above, which may be expected to significantly interfere with the metabolism or excretion of risperidone and/or 9-hydroxyrisperidone, that may be associated with a significant drug interaction with risperidone, or may pose a significant risk to subjects' participation in the study.
* Subjects who have been previously enrolled into the study.
* Subjects who are unable, in the opinion of the Principal Investigator, to comply fully with the study requirements.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse and serious adverse events after a single injection of RBP-7000 | Day 1-Day 85
  Adverse events, serious adverse events, discontinuations due to AEs, local injection site tolerability, vital signs, physical examinations, laboratory results, use of concomitant medications, clinical symptom assessments, 12-lead ECGs
Maximum plasma concentration (Cmax) after a single injection of RBP-7000 | Pre-Dose to 84 days post-dose
  PK parameter will be determined for both risperidone and total risperidone (risperidone + 9-hydroxyrisperidone) at initial burst, secondary peak (if applicable) and overall.
Time of occurrence of Cmax (Tmax) after a single injection of RBP-7000 | Pre-Dose to 84 days post-dose
  PK parameter will be determined for both risperidone and total risperidone (risperidone + 9-hydroxyrisperidone) at initial burst, secondary peak (if applicable) and overall.
Area under the plasma concentration versus time curve (AUC) after a single injection of RBP-7000 | Pre-Dose to 84 days post-dose
  PK parameter will be determined for both risperidone and total risperidone (risperidone + 9-hydroxyrisperidone) at initial burst, secondary peak (if applicable) and overall.
AUC last after a single injection of RBP-7000 | Day 85
  Overall PK parameter will be determined for both risperidone and total risperidone (risperidone + 9-hydroxyrisperidone).
C last | Day 85
  Overall PK parameter will be determined for both risperidone and total risperidone (risperidone + 9-hydroxyrisperidone).
T last | Day 85
  Overall PK parameter will be determined for both risperidone and total risperidone (risperidone + 9-hydroxyrisperidone).
Apparent elimination rate constant (AUC0-∞, λz) | Pre-dose to 84 days post-dose
  Overall PK parameter will be determined for both risperidone and total risperidone (risperidone + 9-hydroxyrisperidone).
Half life (T1/2) | Pre-dose to 84 days post-dose
  Overall PK parameter will be determined for both risperidone and total risperidone (risperidone + 9-hydroxyrisperidone).

SECONDARY OUTCOMES:
Cmax versus RISPERDAL® CONSTA® historical data | Pre-Dose to 84 days post-dose
  The distribution of RBP-7000 compared to those obtained in a previous single-dose study of RISPERDAL® CONSTA®.

CONTACTS AND LOCATIONS:
Locations (1):
- CRI Worldwide, Willingboro, New Jersey, United States